CLINICAL TRIAL: NCT05666999
Title: Post-market Clinical Follow-up Study for a CE Marked Wound Care Product (FibDex®) to Compare the Clinical Performance and Safety in it's Established Intended Use of Split Thickness Skin Graft Donor Site Wounds
Brief Title: Post-market Clinical Follow-up Study for a CE Marked Wound Care Product (FibDex®)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: UPM Kymmene Oyj announced on April 2, 2025, the closure of Biomedicals business. As a result, FibDex manufacturing and sales will discontinue. The premature termination is due to business decision, not related to any safety concerns of FibDex.
Sponsor: UPM-Kymmene Corporation (Industry)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FibDex 2-2022
Record Dates: First submitted 2022-09-12; First posted 2022-12-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Skin Transplantation
Keywords: Skin Transplantation; Donor site; STSG; FibDex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects will be randomized by using a sealed envelope system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FibDex (Other): IMD
  Interventions: Device: FibDex®
- Suprathel (Active Comparator): Primary Comparator.
  Interventions: Device: Suprathel
- Aquacel Foam (Active Comparator): Secondary Comparator.
  Interventions: Device: Aquacel Foam

INTERVENTIONS:
Device: FibDex® — To monitor and compare the clinical performance and safety of the CE marked wound care product (FibDex®) when used according to its intended use for patients or individuals with split thickness skin graft (STSG) donor site wounds.
  Arms: FibDex
Device: Suprathel — To monitor and compare the clinical performance and safety of the CE marked wound care product (FibDex®) when used according to its intended use for patients or individuals with split thickness skin graft (STSG) donor site wounds.
  Arms: Suprathel
Device: Aquacel Foam — To monitor and compare the clinical performance and safety of the CE marked wound care product (FibDex®) when used according to its intended use for patients or individuals with split thickness skin graft (STSG) donor site wounds.
  Arms: Aquacel Foam

SUMMARY:
FibDex® 2-2022 is a sponsored, post-marketing clinical follow-up (PMCF) study to monitor the clinical performance and safety of the CE marked product nanofibrillar cellulose (NFC) wound dressing, FibDex®, when used according to its intended use for patients or individuals with split thickness skin graft (STSG) donor site wounds and to compare clinical performance and safety of FibDex® to current clinical practice.

DETAILED DESCRIPTION:
STSG is a reconstructive procedure that is most used for management of burn injuries. Skin harvesting creates a new partial thickness wound, a donor site that causes additional pain for the patient during the postoperative recovery. Therefore, and because wound healing complications, such as delayed healing and infections, are common donor sites, the donor sites are problematic to treat. A dressing that wound provide optimal healing, low costs, and minimal pain with few dressing changes would be a preferred choice for treatment of donor sites. NFC wound dress, like FibDex, are used for providing these kinds of benefits to patients and better healing result.

This is a sponsored prospective, randomized, controlled, non-blinded, non-inferiority study. Subjects will be treated with the IMD or the comparator and act as their own controls. Subjects will be followed up for up to POD 365. Purpose of this PMCF study for FibDex is to gather data for updating the clinical evaluation and assess if new data gained over time has a bearing on the risk-benefit assessment or if there are some needs to make changes to the product or the package. Clinical evaluation is ongoing and happens throughout the medical devices lifetime. Clinical safety need to be analyzed periodically according to MDR requirements. For class IIb products, like FibDex, it means clinical safety update every year. This study is part of that evaluation.

Aim is to get 48 randomized STSG wounds. Study methods during this study are using the IMD or the comparator after the surgery, subject diaries, pain questionnaires, scar quality assessments by investigator and study subjects and visual observation by the delegated site staff. Also, photos of the healing process will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged at least 18 years when signing the informed consent
2. Subjects with wounds that need split thickness skin grafting (STSG)
3. Subjects that have at least one STSG donor site wound at least 5 x 5 cm and maximum 20 x 30 cm or two STSG donor site wounds of same size, at least 5 x 5 cm and maximum 20 x 30 cm, anatomically close to each other or on anatomically similar area in the opposite extremity or body area.

Exclusion Criteria:

1. Subjects allergic to, or have had an allergic reaction to IMDs components (wood cellulose and polypropylene) or the comparator's components (polylactic acid-based copolymer or natrium carboxymethylcellulose)
2. Pregnant or breast-feeding women
3. Subjects with solid organ transplantation
4. Any other medical condition, compliance, or medication according to Investigator ́s evaluation considered as justified reason for exclusion
5. Vulnerable subject (such as retarded person, person in nursing home, prisoner, patient in emergency)
6. STSG donor site wound(s) on sensitive skin areas, such as the facial area, the genital area or mucous membranes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Wound healing | Post operative day 21
  Wound healing percentage (%) is evaluated by the investigator on POD 21 by removing the dressing and assessing the epithelization.
Wound healing | between post operative day 28-42, if not healed in 3 weeks
  Wound healing percentage (%) is evaluated by the investigator

SECONDARY OUTCOMES:
Subject pain | Diary for post operative days 0 to 21, NRS-scale 1 year.
  Using a patient diary and NRS scale 0-10 (0= no pain,10= worst pain ever)
Epithelialization percentage | post operative day 21
  healing process evaluated by the investigator
Scar quality | day 365
  quality of the scar evaluated by patient
Scar quality | 1 year
  quality of the scar evaluated by observer (investigator)
Adverse events | 1 year
  Total number of adverse events and device defects
Workload during the study visits | Post operative day 21
  To monitor the workload needed e.g. number of extra dressings before post operative day 21 evaluation by using case report forms
Safety of Investigational material | post operative day 21
  Number of IMD or comparator related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kari Luukko, Dr.Tech, Study Director — Director, Quality Assurance
Locations (1):
- Helsinki University Hospital, Espoo, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No